CLINICAL TRIAL: NCT05041660
Title: Using Virtual Reality and Sensor Technology to Enhance Outcomes From Treatment for Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Drexel Coulter Translational Research Partnership Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1906007227
Record Dates: First submitted 2019-10-22; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Binge Eating; Inhibition (Psychology)
Keywords: Inhibitory control; Virtual reality; Binge eating; Continuous glucose monitoring
MeSH Terms: conditions — Bulimia; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: The study is a 2x2 factorial design with the factors being VR (VR/non-VR) and ICT (ICT/Sham).
Who Masked: Participant
Masking Description: Participants and investigators will not be aware who is receiving the sham ICT and who is receiving the real ICT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VR ICT (Experimental): Virtual-reality-based inhibitory control training done daily at home for 6 weeks.
  Interventions: Other: Virtual-reality-based training; Other: Inhibitory Control Training
- VR Sham ICT (Sham Comparator): Virtual-reality-based sham inhibitory control training (i.e., one that does not include a "stop" signal and that thus does not truly train inhibitory control) done daily at home for 6 weeks.
  Interventions: Other: Virtual-reality-based training; Other: Sham Inhibitory Control Training
- Non-VR ICT (Active Comparator): Computerized inhibitory control training done daily at home for 6 weeks.
  Interventions: Other: Inhibitory Control Training; Other: Computerized training
- Non-VR Sham ICT (Sham Comparator): Computerized sham inhibitory control training (i.e., one that does not include a "stop" signal and that thus does not truly train inhibitory control) done daily at home for 6 weeks.
  Interventions: Other: Sham Inhibitory Control Training; Other: Computerized training

INTERVENTIONS:
Other: Virtual-reality-based training — Uses virtual reality for the inhibitory control training, rather than a relatively simplistic computerized training.
  Other Names: VR
  Arms: VR ICT; VR Sham ICT
Other: Inhibitory Control Training — Uses an active inhibitory control training which includes a "stop" signal.
  Other Names: ICT
  Arms: Non-VR ICT; VR ICT
Other: Sham Inhibitory Control Training — Uses an inhibitory control training which does not include a "stop" signal.
  Arms: Non-VR Sham ICT; VR Sham ICT
Other: Computerized training — Uses a relatively simplistic computerized training.
  Arms: Non-VR ICT; Non-VR Sham ICT

SUMMARY:
This study evaluates whether virtual-reality-based inhibitory control trainings are more effective than computerized trainings in reducing binge eating symptomatology. These trainings are used to improve people's ability to resist their impulses towards highly palatable foods (such as chips or cookies). These trainings also offer promise as a companion to Cognitive Behavioral Therapy, an often used and relatively effective therapeutic methodology.

DETAILED DESCRIPTION:
Low levels of inhibitory control (i.e., the ability to withhold a quick, automatic response) is strongly linked with binge eating pathology. One of the most widely used and effective treatments for binge eating leaves 40-60% of patients partially or fully symptomatic at post-treatment. Researchers have begun to investigate the efficacy of computerized inhibitory control trainings (ICTs), which are tasks in which participants are asked repeatedly withhold a keypress responses to food stimuli. The intention of these trainings is to improve inhibitory control and to, in turn, reduce dysregulated eating behavior.

Results for the efficacy of ICTs are promising, yet mixed. ICTs that are gamified (i.e., turned into a video game) using virtual reality technology have high potential to address the barriers which may be limiting the efficacy of previous ICTs. The current study aims to finalize development and test the feasibility, acceptability and preliminary efficacy of the first-ever virtual reality ICT (VR-ICT) for individuals with binge eating pathology.

Thus, the study's aims are as follows:

Primary aim 1: Enhance features of a previously developed, VR-based ICT for binge eating.

Primary aim 2: Examine the feasibility and acceptability of the VR ICT training program.

Primary aim 3: Examine the efficacy of VR-ICT versus a non-VR ICT and ICT vs. sham training, for reductions in binge eating from pre to post-treatment and at follow-up.

Based on previous research and data from a pilot study, the investigators hypothesize a) that the VR ICT training program will be feasible and acceptable and b) that the VR-ICT and ICT will produce superior reductions in binge eating from pre- to post-treatment and at follow-up, as compared, respectively, with the non-VR ICT and the sham ICT.

ELIGIBILITY:
Inclusion Criteria:

* Speak, write, and understand English
* Age 18-65 years
* Experience objectively or subjectively large binge eating episodes once per week or more for the past three months

  * Objectively large binge episodes are defined by the Eating Disorder Examination (EDE; a measure employed in this study) as consisting of at least two full meals of two courses at each (i.e., four courses total) or of at least three main courses
  * Participants, also as per the EDE, must also experience a loss of control over their eating for the given episode to qualify as an objective binge
  * Subjective binges are those which do not meet the food quantity criteria but during which participants experience a loss of control and feel they have eaten too much
* If applicable, have stable psychiatric medication for the past three months.

Exclusion Criteria:

* Acute suicide risk
* Are planning on receiving psychological treatment for binge eating during the course of their participation in the study
* Are planning to participate in a structured weight loss treatment program (e.g., WeightWatchers, behavioral weight loss treatment) during the course of their participation in the study
* Are currently receiving weight loss treatment
* Have a BMI below 17.5
* Co-morbid clinically significant psychological disorder that would require attention beyond the study treatment (i.e., bipolar I disorder, substance dependence, and/or psychotic conditions)
* Diagnosis of intellectual disability or autism spectrum disorder
* History of neurological condition or traumatic brain injury
* Current pregnancy or intention to become pregnant during the course of their participation
* History of bariatric surgery
* Are currently using a stimulant medication (e.g., Ritalin, Adderall)
* No internet connection at home

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Protocol recruitment | The investigators will assess adherence at follow-up assessments (18 weeks after baseline assessment)
  This outcome will be assessed according to whether the investigators can recruit at least 40 participants. This forms the first half of the assessment of the protocol's feasibility.
Protocol retention | The investigators will assess adherence at follow-up assessments (18 weeks after baseline assessment)
  This outcome will be assessed according to whether > 75% of participants completed all assessments. This forms the second half of the assessment of the protocol's feasibility.
Protocol adherence | The investigators will assess adherence at follow-up assessments (18 weeks after baseline assessment).
  This outcome will be assessed according to whether participants completed ≥ 75% of all daily training sessions. This forms the first half of the assessment of the protocol's acceptability.
Protocol satisfaction | The investigators will assess satisfaction at follow-up assessments (18 weeks after baseline assessment).
  This outcome will be assessed according to whether the average participant rating is >= 4 on all questions on the Technology Reactions and Acceptance and Technology Expectancy Questionnaires. This forms the second half of the assessment of the protocol's acceptability.
Impact of VR + ICT vs. VR + Sham on binge eating frequency | The investigators will assess efficacy at post-treatment (6 weeks after baseline) and at follow-up (18 weeks after baseline).
  This outcome will be assessed according to whether participation in the VR + ICT condition produces a larger change in binge eating episodes than does participation in the VR + Sham condition, as measured using the binge module of the Eating Disorder Examination version 17.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Manasse, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Drexel Universitty, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No